CLINICAL TRIAL: NCT03777852
Title: Emotional Evaluation and Reconstructed Breast Satisfaction After Breast Cancer Treatment: Breast Q Questionary
Brief Title: Emotional Evaluation and Reconstructed Breast Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Helio Carrara, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Juçara Phd Thesis; Helio Carrara (Other: DGO-FMRP-USP)
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-12

CONDITIONS: Malignant Neoplasm of the Breast
Keywords: breast cancer, breast surgery, breast reconstruction,
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A group of women will be evaluated twice, being one before the intervention and the second after the breast cancer reconstruction surgery
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-surgery First Breast Q (Experimental): Women with proven breast cancer diagnosis. Respond to the First Breast Q questionnaire..
  Interventions: Diagnostic Test: First Questionnaire application
- Post-surgery Second Breast Q (Active Comparator): The Second Breast Q questionnaire will be applied to this group that will be composed of the women of the first group submitted to reconstructive breast cancer surgery.
  Interventions: Diagnostic Test: Second Questionnaire application

INTERVENTIONS:
Diagnostic Test: First Questionnaire application — Women with breast cancer will respond to the First Breast Q questionnaire before treatment with breast cancer reconstruction surgery.
  Other Names: First Breast Q questionnaire
  Arms: Pre-surgery First Breast Q
Diagnostic Test: Second Questionnaire application — Women with breast cancer will respond to the Second Breast Q questionnaire after treatment with breast cancer reconstruction surgery.
  Other Names: Post reconstruction breast cancer
  Arms: Post-surgery Second Breast Q

SUMMARY:
Data from the National Cancer Institute (Inca) reveal that breast cancer is the most common type of cancer among women worldwide. In Brazil, it is second only to non-melanoma skin cancer. Breast cancer is a feared disease in the female universe because it is considered one of the major causes of death due to neoplasia among women. It brings also the stigma of suffering, mutilation, loss of female identity and loss of body contour. Among other issues, problems with body self-image may have an impact on sexuality and fertility, and also, the incapacity to breastfeed. Breast reconstruction can restore the patient's shape and physical integrity, among other benefits. The research justifies itself because information about the satisfaction of breast reconstruction can be achieved. It is also known that women having breast reconstruction after a mastectomy due to cancer have a favorable evolution. This study will analyze body contour satisfaction of women undergoing mastectomy and breast reconstruction as part of their breast cancer treatment. The Breast Q questionnaire will be used to measure patients satisfaction.

DETAILED DESCRIPTION:
This is a prospective, quasi-experimental study. The subject sample will be composed of women submitted to mastectomy due to breast cancer and to breast reconstruction as part of their treatment. They will be evaluated twice. One when they receive the cancer diagnosis and the other six months after de reconstruction surgery. On both occasions, they will answer the Brest Q questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* women over eighteen years of age;
* women with proven histological diagnosis of breast cancer;
* women who have an indication of mastectomy as part of their treatment;
* women who have breast reconstruction, regardless of the technique used, as part of their treatment;
* women under 70 years of age at the time of the reconstructive surgery

Exclusion Criteria:

* women diagnosed with breast cancer and treated with conservative surgeries;
* women who refuse reconstruction as part of treatment;
* women who refused surgery as part of the treatment for breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Post-treatment Satisfaction | Six month
  Comparison of results between the first and the second Breast Q score. This score represents questionnaries about diferents domains and each question has four possible dimensions. The values of these dimensions varies from 1 to 4 (Likert Scale). The sum of each domain raw score scale will be plotted in the Breast Q Conversion Table to convert the summed domain score to a Equivalent Rasch Transformed Score with values ranging from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Helio HA Carrara, MD, PhD, Principal Investigator — Gynecology & Obstetrics Departament, Ribeirão Preto Medical School, USP.
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen WA, Mundy LR, Ballard TN, Klassen A, Cano SJ, Browne J, Pusic AL. The BREAST-Q in surgical research: A review of the literature 2009-2015. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):149-62. doi: 10.1016/j.bjps.2015.11.013. Epub 2015 Nov 26. PMID 26740288
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Mundy LR, Homa K, Klassen AF, Pusic AL, Kerrigan CL. Breast Cancer and Reconstruction: Normative Data for Interpreting the BREAST-Q. Plast Reconstr Surg. 2017 May;139(5):1046e-1055e. doi: 10.1097/PRS.0000000000003241. PMID 28445351
- [Background] Payne RM, Siotos C, Manahan MA, Rosson GD, Cooney CM. Breast Cancer and Reconstruction: Normative Data for Interpreting the BREAST-Q. Plast Reconstr Surg. 2018 Jan;141(1):180e-181e. doi: 10.1097/PRS.0000000000003970. No abstract available. PMID 28938344
- [Background] Saiga M, Taira N, Kimata Y, Watanabe S, Mukai Y, Shimozuma K, Mizoo T, Nogami T, Iwamoto T, Motoki T, Shien T, Matsuoka J, Doihara H. Development of a Japanese version of the BREAST-Q and the traditional psychometric test of the mastectomy module for the assessment of HRQOL and patient satisfaction following breast surgery. Breast Cancer. 2017 Mar;24(2):288-298. doi: 10.1007/s12282-016-0703-6. Epub 2016 May 14. PMID 27179527
- [Background] Fuzesi S, Cano SJ, Klassen AF, Atisha D, Pusic AL. Validation of the electronic version of the BREAST-Q in the army of women study. Breast. 2017 Jun;33:44-49. doi: 10.1016/j.breast.2017.02.015. Epub 2017 Mar 7. PMID 28279888